CLINICAL TRIAL: NCT07096752
Title: Screening and Validation of Serum Protein Biomarkers for Early Diagnosis of Gastric Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Hao-Jie Li, Doctor, Shanghai Zhongshan Hospital
Other Study IDs: B2025-308R
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer (Diagnosis)
MeSH Terms: conditions — Stomach Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric cancer: Patients with histopathologically confirmed gastric cancer
- Non Gastric Cancer: Healthy controls or patients with histologically confirmed precancerous gastric lesions that have not yet progressed to malignancy.

SUMMARY:
This study focuses on the discovery of protein biomarkers for the early diagnosis of gastric cancer and the development of corresponding detection methods. By employing advanced mass spectrometry-based proteomic technologies, the investigators conducted an in-depth analysis of a large cohort of clinical samples to identify specific protein biomarkers capable of accurately distinguishing gastric cancer patients from healthy individuals. The findings from this research are expected to facilitate the development of novel non-invasive or minimally invasive diagnostic approaches, thereby improving early detection, enhancing patient prognosis, and increasing survival rates.

ELIGIBILITY:
Inclusion Criteria

Gastric cancer patients enrolled in this study must meet all of the following criteria:

1. Male or female, aged ≥18 and ≤95 years.
2. Histopathologically confirmed gastric cancer, as defined by the 2024 edition of the Chinese Society of Clinical Oncology (CSCO) Guidelines for the Diagnosis and Treatment of Gastric Cancer.
3. No prior anti-tumor treatment (including radiotherapy, chemotherapy, targeted therapy, or immunotherapy).
4. Availability of complete clinicopathological data and follow-up information.

Patients with precancerous gastric lesions must meet all of the following criteria:

1. Male or female, aged ≥18 and ≤95 years.
2. Histopathologically confirmed absence of gastric cancer.
3. Diagnosis consistent with precancerous gastric lesions as defined by the American Society for Gastrointestinal Endoscopy (ASGE, 2015 edition).
4. Availability of complete clinicopathological data and follow-up information.

Healthy controls must meet all of the following criteria:

1. Male or female, aged ≥18 and ≤95 years.
2. Histopathologically confirmed absence of gastric cancer.
3. No evidence of precancerous gastric lesions.
4. Availability of complete clinicopathological data and follow-up information.

Exclusion Criteria

Patients meeting any of the following conditions will be excluded:

1. History of prior malignancy or cancer treatment.
2. Presence of concurrent malignancies of other types.
3. Inability to tolerate gastroscopy.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study recruits two main populations: patients with gastric cancer and non-gastric cancer participants. The latter group includes two subgroups: individuals with precancerous gastric lesions and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance of the Serum Protein Biomarker-Based Model for Gastric Cancer | 3 years
  Evaluation of the sensitivity and specificity of a diagnostic model constructed using key serum protein biomarkers for the early detection of gastric cancer.

SECONDARY OUTCOMES:
Predictive performance of the serum protein model for the progression risk from precancerous gastric lesions to gastric cancer | 3 years
  Predictive performance of the serum protein model for the progression risk from precancerous gastric lesions to gastric cancer, evaluated by prediction accuracy and area under the ROC curve (AUC).
Predictive performance of the serum protein model for response to neoadjuvant therapy in gastric cancer | 3 years
  Predictive performance of the serum protein model for response to neoadjuvant therapy in gastric cancer, assessed by prediction accuracy and AUC.
Prognostic performance of the serum protein model in gastric cancer patients | 3 years
  Prognostic performance of the serum protein model in gastric cancer patients, measured by prediction accuracy and AUC.

IPD SHARING:
Plan to Share IPD: No